CLINICAL TRIAL: NCT04613193
Title: Blood Pressure Reduction in Patients With Asymptomatic Aortic VALVE Stenosis
Acronym: BP-AVALVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henrik Wiggers (Other)
Collaborators: Danish Heart Foundation (Other)
Responsible Party: Sponsor-Investigator, Henrik Wiggers, Consultant, Associate professor, MD, PhD, DMSc, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BP-AVALVE
Record Dates: First submitted 2020-07-09; First posted 2020-11-03 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Aortic Valve Stenosis; Hypertension,Essential; Heart Failure
Keywords: Aortic Valve Stenosis; Hypertension; Heart failure
MeSH Terms: conditions — Aortic Valve Stenosis; Essential Hypertension; Heart Failure; Hypertension

STUDY DESIGN:
Intervention Model Description: 1. BP-AVALVE I: 60 patients will be randomized (1:1) to either strict BP control (N=30) or conventional treatment (N=30). Treatment period will be 12 months.
  2. BP-AVALVE II: 200 patients will be randomized (1:1) to either strict BP control as in study 1 (N=100) or conventional care as in study 1 (N=100). Average treatment period will be 2 (1-3) years.
  3. BP-AVALVE III: Patients from BP-AVALVE-II continue in the randomized design until they develop symptoms of AS or have been followed for 10 (7-13) years. Patients will be reexamined at the end of the study period or in case they develop symptoms or LV failure and thus indication of valve replacement.
  Since the medicinal products used in this study is not the subject of the trial, the Danish Medicines Agency has classified this study as a clinical trial, in which medicinal products are used as a tool to induce a well-known physiological response. Therefor no further approval from the Danish Medicine Agency is required.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strict BP intervention group (Active Comparator): SBP < 120 mmHg and a reduction in SBP of >= 15 mmHg
  Interventions: Other: Blood presssure reduction
- Conventional BP control group (Other): In patients < 75 years: SBP = 135 mmHg In patients >/= 75 years: SBP = 145 mmHg
  Interventions: Other: Blood presssure reduction

INTERVENTIONS:
Other: Blood presssure reduction — Patients will be uptitrated in antihypertensive treatment until the treatment target is achieved.

SUMMARY:
The aim of this study is to investigate the effect of strict blood pressure control versus conventional care in patients with asymptomatic moderate to severe aortic valve stenosis.

The study is a randomized (1:1), open label, controlled intervention trial.

Hypothesis:

1. Strict BP control for 12 months reduces the progression of LV remodelling compared to conventional treatment.
2. Strict BP control for 2 years reduces the increase in aortic valve calcification and LV remodelling compared to conventional treatment.
3. Strict BP reduction for up to 10 years reduces the need for aortic valve replacement and cardiovascular events compared to conventional care.

ELIGIBILITY:
Inclusion Criteria:

* Aortic valve peak velocity (Vmax) of 3.0-5.0 m/s and/or aortic valve area (AVA) ≤ 1.2 cm2
* Blood pressure: SBP >= 127 mmHg measured by BP-TRU
* LVEF ≥ 50%
* Age > 18 years
* Safe birth control management (intrauterine devices or hormonal contraceptives (contraceptive pills, implants, transdermal patches, hormonal vaginal devices or injections with prolonged release)) for women of childbearing potential.
* Negative urine-HCG for women of childbearing potential
* Ability to understand the written patient information and to give informed consent.

Exclusion Criteria:

* Symptoms due to AS
* Symptomatic orthostatic hypotension and/or one minute standing SBP < 110 mmHg (16).
* Suspicion of secondary hypertension
* Participation in other randomized drug study (device studies accepted)
* Moderat to severe aortic valve regurgitation e.g. vena contracta > 5 mm, assessed by echocardiography)
* Known or suspected ischemic heart disease (coronary angiography with >70% stenosis in a major epicardial vessel, symptoms or signs of myocardial ischemia, e.g. angina pectoris, wall motion abnormalities). Patients who have previously undergone complete revascularization of major coronary arteries due to angina pectoris are eligible for inclusion.
* Significant coronary obstructive lesions detected by baseline Cardiac CT that requires a revascularisation procedure.
* eGFR < 30 ml/min or end-stage renal disease
* Other disease, comorbidity or treatment making the subject unsuitable for study participation as judged by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2031-01-01 (Estimated); Study Completion 2031-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in LV mass | Changes will be evaluated after an expected average of 12 months treatment
  LV mass as measured by cardiac MR
Change in aortic valve CT calcium volume and aortic peak gradient | Changes will be evaluated after an expected average of 2-3 years treatment
  Cardiac CT and Echocardiography
Clinical composite endpoint: | Will be evaluated after an expected average of 7-13 years of treatment
  Major cardiovascular events including death from cardiovascular causes, aortic valve replacement, non-fatal myocardial infarction, hospitalization for unstable angina pectoris, heart failure, coronary artery bypass surgery, percutaneous coronary intervention, and haemorrhagic and non-haemorrhagic stroke, new onset atrial fibrillation.

SECONDARY OUTCOMES:
LV mass-cavity ratio. | Through study completion, an average of 1 year
  Cardiac MR
LV myocardial fibrosis | Through study completion, an average of 1 year
  Cardiac MR
Myocardial perfusion during rest and stress | Through study completion, an average of 1 year
  Cardiac MR
Aortic peak and mean gradients | Through study completion, an average of 1 year
  Echocardiography
Aortic valve area | Through study completion, an average of 1 year
  Echocardiography
Left ventricular global longitudinal strain | Through study completion, an average of 1 year
  Echocardiography
Valvolu-arterial impedance | Through study completion, an average of 1 year
  Echocardiography
NT-proBNP | Baseline and follow-up
  Blood test
Minnesota living with heart failure questionnaire | Through study completion, an average of 1 year
  Questionnaire
Ambulatory 24-hour blood pressure measurement | Through study completion, an average of 1 year
  Ambulatory 24-hour blood pressure measurement
Dimensions and aortic calcium score of the thoracic aorta. | Through study completion, an average of 2 years
  cardiac CT

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Wiggers, Principal Investigator — Aarhus University Hospital, Department of Cardiology
Locations (6):
- Denmark (6):
  - Dept. of Cardiology, Aarhus University Hospital, Palle Juul-Jensens Boulevard 99, Aarhus
  - Dept. of Cardiology, Herning Hospital, Herning
  - Dept. of cardiology, Horsens Hospital, Horsens
  - Dept. of cardiology, Randers Hospital, Randers
  - Silkeborg Hospital, Silkeborg
  - Dept. of cardiology, Viborg Hospital, Viborg

IPD SHARING:
Plan to Share IPD: No